CLINICAL TRIAL: NCT03020615
Title: Hydroxyurea Management in Kids: Intensive Versus Stable Dosage Strategies
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: St. Jude Children's Research Hospital (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HUGKISS; R34HL127162 (NIH)
Record Dates: First submitted 2017-01-11; First posted 2017-01-13 (Estimated); Results first posted 2021-06-25 (Actual); Last update posted 2021-06-25 (Actual); Status verified 2021-05

CONDITIONS: Sickle Cell Anemia
Keywords: Sickle cell; Hydroxyurea; Infants
MeSH Terms: conditions — Anemia, Sickle Cell | interventions — Hydroxyurea

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Stable Dosing (Active Comparator): In the first 8 weeks (± 2 weeks) of this study, participants will receive standard treatment [a fixed dose of 20 (± 2.5) mg/kg/day of hydroxyurea]. After 8 weeks (± 2 weeks) of standard treatment, participants will be randomized (like flipping a coin) to one of two treatment groups. Group 1 (Stable Dosing) continues standard treatment.
  Interventions: Drug: Hydroxyurea
- Intensive Dosing (Experimental): In the first 8 weeks (± 2 weeks) of this study, participants will receive standard treatment [a fixed dose of 20 (± 2.5) mg/kg/day of hydroxyurea]. After 8 weeks (± 2 weeks) of standard treatment, participants will be randomized (like flipping a coin) to one of two treatment groups. Group 2 (Intensive Dosing) will have their HU dose increased by 5 mg/kg/day every 8 weeks up to a maximum of 35 mg/kg/day.
  Interventions: Drug: Hydroxyurea

INTERVENTIONS:
Drug: Hydroxyurea — Given orally once daily.
  Other Names: HU

SUMMARY:
This is a pilot study, single-blind, randomized, multicenter, therapeutic clinical trial designed to evaluate the feasibility of enrolling infants and toddlers (9 months to 36 months) with sickle cell anemia (SCA; HbSS or HbSβ^0thalassemia), regardless of disease severity, to a therapeutic trial. A prior clinical trial at St. Jude Children's Research Hospital (SJCRH) (BABYHUG, NCT01783990) demonstrated that a fixed dose (20 mg/kg/day) of hydroxyurea was safe and effective in decreasing SCA-related complications in very young children (9-18 months), and largely due to these findings, hydroxyurea is recommended to be offered to all children (≥9 months old) with SCA, independent of disease severity. Nevertheless, children in the treatment arm of BABYHUG continued to experience vaso-occlusive symptoms and to incur organ damage. In clinical trials of older children with SCA, intensification of hydroxyurea to a maximum tolerated dosage (MTD), defined by mild to moderate myelosuppression, may be associated with improved laboratory parameters compared to fixed lower-dosing, but the clinical benefits gained from dose intensification have not been described. Therefore, in this trial, children in the standard treatment arm will receive a fixed dose of hydroxyurea (20 mg/kg/day), and participants in the experimental arm will receive hydroxyurea intensified to MTD, defined by a goal absolute neutrophil count (ANC) of 1500-3000 cells/µL. This trial aims to establish a multicenter infrastructure that will identify, enroll and randomize very young children (9-36 months) to receive fixed dose versus intensified-dose hydroxyurea in a single blinded manner, and to obtain prospective pilot data comparing the clinical and laboratory outcomes between the treatment arms to facilitate design of a definitive phase III trial.

DETAILED DESCRIPTION:
All participants will initially receive hydroxyurea at a dose of ~20 mg/kg/day in an open label fashion for eight weeks (± 2 weeks) prior to randomization. Participants will receive monthly medical evaluations (every 4 ± 2 weeks) where they will have height and weight measurements, medical history, physical examination, and medication adherence assessments. During these monthly visits complete blood counts with absolute reticulocyte count will be monitored. Hemoglobin electrophoresis, complete serum chemistries, urinalysis, lactate dehydrogenase and quality of life measurements will be obtained every 20 (±2) weeks. Transcranial Doppler (TCD) ultrasound velocities will be obtained at study entry (in participants ≥2 years of age) and study exit. Participants randomized to receive hydroxyurea at MTD will have their dose increased by 5 mg/kg/day every 8 weeks, in the absence of toxicity, until a goal ANC of 1500-3000 cells/µL is achieved, up to a maximum of 35 mg/kg/day.

Both groups will receive their assigned treatment for 48 weeks (± 3 weeks). Participants will be in the study for a total of 56 weeks (± 3 weeks) and have 14 clinic visits to the St. Jude outpatient Hematology Clinic during that time. After the 56 weeks, participants will be followed for an additional 30 days for side effects and will then be taken off study.

ELIGIBILITY:
Inclusion Criteria:

* Children with HbSS or sickle hemoglobin (HbS)/β^0thalassemia
* ≥9 to ≤ 36 months of age at study initiation
* Enrollment will occur irrespective of clinical severity

Exclusion Criteria:

Permanent:

* Receiving chronic red blood cell transfusion therapy.
* Condition or chronic illness, which in the opinion of the PI makes participation unsafe.

Transient (participants may be re-evaluated after ≥14 days):

* Recent (<30 days) participation in another clinical intervention trial utilizing an investigational new drug/investigational device exemption (IND/IDE) agent.
* Erythrocyte transfusion in the past 2 months.
* Laboratory Assessments:

  * Hemoglobin <6.0 g/dL
  * Absolute reticulocyte count <80 * 10^3/µL if hemoglobin <9.0 mg/dL
  * Absolute neutrophil count <1.5 * 10^3/µL
  * Platelet count <100 * 10^3/µL
  * Serum creatinine > twice the upper limit of normal for age
  * Alanine aminotransferase (ALT) > twice the upper limit of normal

Ages: 9 Months to 36 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 58 (Actual)
Dates: Start 2017-05-12 (Actual); Primary Completion 2020-06-08 (Actual); Study Completion 2020-06-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeremie Estepp, MD, Principal Investigator — St. Jude Children's Research Hospital
Locations (4):
- United States (4):
  - Emory University/Children's Health Care of Atlanta, Atlanta, Georgia
  - University of Mississippi Medical Center, Jackson, Mississippi
  - St. Jude Children's Research Hospital, Memphis, Tennessee
  - University of Texas Southwestern Medical Center at Dallas, Dallas, Texas

REFERENCES:
- See also: St. Jude Children's Research Hospital — http://www.stjude.org
- See also: Clinical Trials Open at St. Jude — http://www.stjude.org/protocols

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study planned to enroll up to 65 children with sickle cell anemia (SCA) to get 50 randomized in a 27-month period. All eligible participants who consented were enrolled on the study. The duration of the study is based on sample size of 50 patients randomized and/or 27-month period, whichever comes first. Actual recruitment occurred 5/3/2017 to 6/3/2019 and 58 subjects were enrolled to yield 51 randomized at 4 clinical centers.
Pre-assignment Details: Participants without toxicity or with toxicity which requires discontinuation of hydroxyurea (HU) but resolved and participant continuing HU during those eight weeks (±2 weeks), were randomized to receive standard or intensive therapy based on a block randomization (block size of 4 used in each stratum) stratified by clinical center and by baseline age of the participant (9 to <24 months and 24 to 36 months) because of the natural physiologic decline of HbF with increasing age.
Groups:
- Non-Randomized: Participants who came off study prior to randomization
Period: Overall Study
Arm/Group | Stable Dosing | Intensive Dosing | Non-Randomized
Started | 26 | 25 | 7
Completed | 19 | 23 | 0
Not Completed | 7 | 2 | 7
Not completed — Physician Decision | 3 | 1 | 2
Not completed — Parent/guardian/patient choice | 3 | 0 | 4
Not completed — Screen failure | 0 | 0 | 1
Not completed — Death | 1 | 0 | 0
Not completed — Lost to Follow-up | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Non-Randomized Patients: Patients who came off study prior to randomization
- Total: Total of all reporting groups
Arm/Group | Stable Dosing | Intensive Dosing | Non-Randomized Patients | Total
Number analyzed (Participants) | 26 | 25 | 7 | 58
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 26 | 25 | 7 | 58
  Between 18 and 65 years | 0 | 0 | 0 | 0
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Median (Full Range); unit: months] | 9 [9 to 36] | 10 [9 to 32] | 18 [10 to 23] | 10 [9 to 36]
Age, Continuous [Mean (Standard Deviation); unit: months] | 12.9 (7.9) | 12.8 (6.2) | 18.1 (4.7) | 13.5 (7.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 8 | 2 | 25
  Male | 11 | 17 | 5 | 33
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black | 25 | 25 | 6 | 56
  White | 1 | 0 | 0 | 1
  Unknown | 0 | 0 | 1 | 1
  Non-Spanish speaking Non Hispanic | 26 | 23 | 6 | 55
  Non-Spanish speaking Non Hispanic (Unknown) | 0 | 2 | 1 | 3
Region of Enrollment [Count of Participants; unit: Participants]
  United States: St. Jude Children's Research Hospital | 16 | 17 | 0 | 33
  United States: Children's Healthcare of Atlanta | 8 | 5 | 4 | 17
  United States: University of Mississippi Medical Center | 1 | 2 | 2 | 5
  United States: University of Texas Southwestern Medical Center | 1 | 1 | 1 | 3

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients Enrolled.
Description: A count of the number of patients enrolled will be provided.
Time Frame: at baseline
Population: 58 subjects enrolled on study. Of those, n=7 came off study prior to randomization (N=2 came off study due to PI discretion, n=4 came off study due to Parent/guardian/patient choice, and n=1 was a screen failure (HBG)). The remaining n=51 were randomized.
Measure: Count of Participants; unit: Participants
Groups:
- All Participants: All Participants enrolled on study.
Arm/Group | All Participants
Number analyzed (Participants) | 58
Participants | 58

2. Primary Outcome: Number of Patients Randomized
Description: A count of the number of patients randomized will be provided.
Time Frame: Eight weeks (± 2 weeks) after study enrollment
Population: Fifty-one were randomized out of the 58 enrolled.
Measure: Count of Participants; unit: Participants
Arm/Group | Stable Dosing | Intensive Dosing
Number analyzed (Participants) | 26 | 25
Participants | 26 | 25

3. Primary Outcome: Number of Randomized Patients With ≥80% Chronic Medication Compliance
Description: Chronic medication compliance is defined based on medication possession ratio (MPR), a measure of the percentage of time that a patient has access to medication. Each participant's MPR is calculated as [(days medication in family's possession/days prescribed medication) * 100].
Time Frame: At completion of therapy, up to 56 weeks after study enrollment
Population: There were 51 subjects randomized to treatment of which 42 completed the protocol therapy. MPR was calculated on the full study period. The n=9 patients that were withdrawn were counted as <80% chronic medical compliance. Of the n=42 patients that completed protocol treatment, n=41 had ≥80% chronic medication compliance.
Measure: Count of Participants; unit: Participants
Groups:
- Randomized Participants: Number of participants randomized.
Arm/Group | Randomized Participants
Number analyzed (Participants) | 51
Participants | 41

4. Primary Outcome: Number of Patients Who Have the % Fetal Hemoglobin (%HbF) Collected at Baseline and at Study Exit
Description: The number of patients who have successfully provided %HbF at baseline and study exit will be provided.
Time Frame: At baseline and at completion of the protocol, up to 56 weeks after study enrollment
Population: N=42 patients completed the protocol therapy and had labs collected at exit visit.
Measure: Number; unit: Participants
Arm/Group | Stable Dosing | Intensive Dosing
Number analyzed (Participants) | 26 | 25
Participants | 19 | 23

5. Secondary Outcome: Frequency by Reason Given for Refusal for Study Participation
Description: Descriptive statistics of count and frequency will be provided for participants who were approached but refused to be enrolled on the study.
Time Frame: Once, at enrollment
Population: n=154 subjects declined to participate in HUGKISS and provided the following reasons for declining to participate.
Measure: Count of Participants; unit: Participants
Groups:
- Subjects Approached Who Declined Participation: Subjects who declined to participate in HUGKISS and provided reasons for declining
Arm/Group | Subjects Approached Who Declined Participation
Number analyzed (Participants) | 154
Participants
  Does not meet eligibility criteria | 33
  Family wants more time to consider participation | 31
  Child on hydroxyurea (HU) | 29
  Unknown reason | 17
  Not interested in HU | 16
  Poor clinic visit compliance | 13
  Not interested in research | 10
  Logistics - travel distance to site, frequency of appointments | 5

6. Secondary Outcome: Number of Patients With Hospitalizations by Arm
Description: The number of patients with hospitalizations will be provided by arm. This analysis approach is different than what was written in the protocol due to small number of participants with hospitalizations and small number of hospitalization events.
Time Frame: From baseline through completion of therapy, up to 56 weeks
Population: The n=51 subjects that were randomized to treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Stable Dosing | Intensive Dosing
Number analyzed (Participants) | 26 | 25
Participants | 2 | 2

7. Secondary Outcome: Cumulative Number of Hospitalizations by Arms
Description: The total number of hospitalization events will be provided by arms. This analysis approach is different than what was written in the protocol due to small number of participants with hospitalizations and small number of hospitalization events.
Time Frame: From baseline through completion of therapy, up to 56 weeks
Population: The n=51 subjects that were randomized to treatment.
Measure: Number; unit: hospitalizations
Arm/Group | Stable Dosing | Intensive Dosing
Number analyzed (Participants) | 26 | 25
hospitalizations | 4 | 5

8. Secondary Outcome: Mean Change in Hemoglobin (g/dL)
Description: Descriptive statistics of the change between baseline and completion of the study will be provided and will be compared between two treatment arms using two sample t-test or exact Wilcoxon Rank Sum test depending on the normality of the data tested by the Shapiro-Wilk test.
Time Frame: From baseline at study entry to completion of therapy, up to 56 weeks
Population: Change calculations require subjects to have values at both baseline and exit visits. N=51 patients were randomized (n=25 to the Intensive arm and n=26 to the standard arm.) N=42 subjects completed protocol therapy (n=23 to the intensive arm and n=19 to the standard arm.) All n=42 that completed the study had HGB measurements at both baseline and at exit visit.
Measure: Mean (Standard Deviation); unit: g/dL
Groups:
- Overall: All subjects who completed protocol therapy
Arm/Group | Stable Dosing | Intensive Dosing | Overall
Number analyzed (Participants) | 19 | 23 | 42
g/dL | 0.42 (0.84) | 1.15 (1.21) | 0.82 (1.11)
Statistical Analysis 1: Comparison: Stable Dosing vs Intensive Dosing; Test type: Superiority; p = 0.033, t-test, 2 sided

9. Secondary Outcome: Median Change in Hemoglobin (g/dL)
Description: Descriptive statistics of the change between baseline and completion of the study will be provided.
Time Frame: From baseline at study entry to completion of therapy, up to 56 weeks
Population: Change calculations require subjects to have values at both baseline and exit visits. N=51 patients were randomized (n=25 to the Intensive arm and n=26 to the standard arm.) N=42 subjects completed protocol therapy (n=23 to the intensive arm and n=19 to the standard arm.) All n=42 that completed the study had hemoglobin (HGB) measurements at both baseline and at exit visit.
Measure: Median (Full Range); unit: g/dL
Arm/Group | Stable Dosing | Intensive Dosing | Overall
Number analyzed (Participants) | 19 | 23 | 42
g/dL | 0.40 [-1.30 to 1.50] | 1.20 [-1.90 to 3.35] | 1.05 [-1.90 to 3.35]

10. Secondary Outcome: Mean Change in Fetal Hemoglobin (%)
Description: Descriptive statistics of the change between baseline and completion of the study will be provided.
Time Frame: From baseline at study entry to completion of therapy, up to 56 weeks
Population: Change calculations require subjects to have values at both baseline and exit visits. N=51 patients were randomized (n=25 to the Intensive arm and n=26 to the standard therapy arm.) N=42 subjects completed protocol therapy (n=23 in the intensive arm and n=19 in the standard arm.) All 42 that completed the study had Hemoglobin F (HbF) measurements at both baseline and at exit visit.
Measure: Mean (Standard Deviation); unit: percentage of Hemoglobin F
Arm/Group | Stable Dosing | Intensive Dosing | Overall
Number analyzed (Participants) | 19 | 23 | 42
percentage of Hemoglobin F | -6.97 (18.97) | 7.67 (12.09) | 1.05 (17.06)

11. Secondary Outcome: Median Change in Fetal Hemoglobin (%)
Description: as for outcome 8
Time Frame: From baseline at study entry to completion of therapy, up to 56 weeks
Population: as for outcome 10
Measure: Median (Full Range); unit: percentage of Hemoglobin F
Arm/Group | Stable Dosing | Intensive Dosing | Overall
Number analyzed (Participants) | 19 | 23 | 42
percentage of Hemoglobin F | 0.20 [-60.70 to 4.80] | 8.00 [-23.50 to 24.70] | 1.70 [-60.70 to 24.70]
Statistical Analysis 1: Comparison: Stable Dosing vs Intensive Dosing; Test type: Superiority; p = 0.0005, Exact Wilcoxon (Mann-Whitley), two-sided

12. Secondary Outcome: Mean Change in Mean Corpuscular Volume (fL)
Description: Descriptive statistics of the change between baseline and completion of the study will be provided.
Time Frame: From baseline at study entry to completion of therapy, up to 56 weeks
Population: Change calculations require subjects to have values at both baseline and exit visits. N=51 patients were randomized (n=25 to the Intensive arm and n=26 to the standard therapy arm.) N=42 subjects completed protocol therapy (n=23 in the intensive arm and n=19 in the standard arm.) All 42 that completed the study had mean corpuscular volume (MCV) measurements at both baseline and exit visits.
Measure: Mean (Standard Deviation); unit: fL
Arm/Group | Stable Dosing | Intensive Dosing | Overall
Number analyzed (Participants) | 19 | 23 | 42
fL | 5.87 (6.17) | 11.36 (4.84) | 8.88 (6.08)

13. Secondary Outcome: Median Change in Mean Corpuscular Volume (fL)
Description: as for outcome 8
Time Frame: From baseline at study entry to completion of therapy, up to 56 weeks
Population: as for outcome 12
Measure: Median (Full Range); unit: fL
Arm/Group | Stable Dosing | Intensive Dosing | Overall
Number analyzed (Participants) | 19 | 23 | 42
fL | 8.00 [-7.10 to 16.00] | 9.60 [5.40 to 20.10] | 8.70 [-7.10 to 20.10]
Statistical Analysis 1: Comparison: Stable Dosing vs Intensive Dosing; Test type: Superiority; p = 0.011, Exact Wilcoxon (Mann-Whitney), two-sided

14. Secondary Outcome: Mean Change in Absolute Reticulocyte Count (*10^3 Reticulocytes/µL)
Description: as for outcome 8
Time Frame: From baseline at study entry to completion of therapy, up to 56 weeks
Population: Change calculations require subjects to have values at both baseline and exit visits. N=51 patients were randomized (n=25 to the Intensive arm and n=26 to the standard therapy arm.) N=42 subjects completed protocol therapy (n=23 in the intensive arm and n=19 in the standard arm.) N=41 of the n=42 subjects that completed the study had absolute reticulocyte count (ARC) measurements at both baseline and exit visits.
Measure: Mean (Standard Deviation); unit: *10^3 reticulocytes/µL
Arm/Group | Stable Dosing | Intensive Dosing | Overall
Number analyzed (Participants) | 19 | 22 | 41
*10^3 reticulocytes/µL | -83.69 (65.65) | -145.43 (107.10) | -116.82 (94.52)
Statistical Analysis 1: Comparison: Stable Dosing vs Intensive Dosing; Test type: Superiority; p = 0.030, t-test, 2 sided

15. Secondary Outcome: Median Change in Absolute Reticulocyte Count (*10^3 Reticulocytes/µL)
Description: Descriptive statistics of the change between baseline and completion of the study will be provided.
Time Frame: From baseline at study entry to completion of therapy, up to 56 weeks
Population: as for outcome 14
Measure: Median (Full Range); unit: *10^3 reticulocytes/µL
Arm/Group | Stable Dosing | Intensive Dosing | Overall
Number analyzed (Participants) | 19 | 22 | 41
*10^3 reticulocytes/µL | -91.6 [-202.3 to 55.1] | -175.9 [-300 to 109.1] | -120.5 [-300 to 109.1]

16. Secondary Outcome: Mean Change in White Blood Cell Count (*10^3 White Blood Cells/µL)
Description: Descriptive statistics of the change between baseline and completion of the study will be provided.
Time Frame: From baseline at study entry to completion of therapy, up to 56 weeks
Population: Change calculations require subjects to have values at both baseline and exit visits. N=51 patients were randomized (n=25 to the Intensive arm and n=26 to the standard therapy arm.) N=42 subjects completed protocol therapy (n=23 in the intensive arm and n=19 in the standard arm.) All 42 that completed the study had white blood cell (WBC) measurements at both baseline and exit visits.
Measure: Mean (Standard Deviation); unit: *10^3 white blood cells/µL
Arm/Group | Stable Dosing | Intensive Dosing | Overall
Number analyzed (Participants) | 19 | 23 | 42
*10^3 white blood cells/µL | -0.32 (4.78) | -5.64 (5.56) | -3.23 (5.81)

17. Secondary Outcome: Median Change in White Blood Cell Count (*10^3 White Blood Cells/µL)
Description: as for outcome 8
Time Frame: From baseline at study entry to completion of therapy, up to 56 weeks
Population: as for outcome 16
Measure: Median (Full Range); unit: *10^3 white blood cells/µL
Arm/Group | Stable Dosing | Intensive Dosing | Overall
Number analyzed (Participants) | 19 | 23 | 42
*10^3 white blood cells/µL | -0.77 [-8.07 to 12.46] | -4.50 [-20.35 to 4.23] | -3.14 [-20.35 to 12.46]
Statistical Analysis 1: Comparison: Stable Dosing vs Intensive Dosing; Test type: Superiority; p = 0.0009, Exact Wilcoxon (Mann-Whitney), two-sided

18. Secondary Outcome: Mean Change in Absolute Neutrophil Count (*10^3 Neutrophils/µL)
Description: Descriptive statistics of the change between baseline and completion of the study will be provided.
Time Frame: From baseline at study entry to completion of therapy, up to 56 weeks
Population: Change calculations require subjects to have values at both baseline and exit visits. N=51 patients were randomized (n=25 to the Intensive arm and n=26 to the standard therapy arm.) N=42 subjects completed protocol therapy (n=23 in the intensive arm and n=19 in the standard arm.) N=41 of the 42 that completed the study had absolute neutrophil count (ANC) measurements at both baseline and exit visits.
Measure: Mean (Standard Deviation); unit: *10^3 neutrophils/µL
Arm/Group | Stable Dosing | Intensive Dosing | Overall
Number analyzed (Participants) | 18 | 23 | 41
*10^3 neutrophils/µL | 0.74 (2.53) | -1.69 (2.09) | -0.62 (2.57)

19. Secondary Outcome: Median Change in Absolute Neutrophil Count (*10^3 Neutrophils/µL)
Description: as for outcome 8
Time Frame: From baseline at study entry to completion of therapy, up to 56 weeks
Population: as for outcome 18
Measure: Median (Full Range); unit: *10^3 neutrophils/µL
Arm/Group | Stable Dosing | Intensive Dosing | Overall
Number analyzed (Participants) | 18 | 23 | 41
*10^3 neutrophils/µL | 0.35 [-2.13 to 9.30] | -1.43 [-8.10 to 1.49] | -0.52 [-8.10 to 9.30]
Statistical Analysis 1: Comparison: Stable Dosing vs Intensive Dosing; Test type: Superiority; p = 0.0004, Exact Wilcoxon (Mann-Whitney), two-sided

20. Secondary Outcome: Mean Change in Platelet Count (*10^3 Platelets/µL)
Description: Descriptive statistics of the change between baseline and completion of the study will be provided.
Time Frame: From baseline at study entry to completion of therapy, up to 56 weeks
Population: Change calculations require subjects to have values at both baseline and exit visits. N=51 patients were randomized (n=25 to the Intensive arm and n=26 to the standard therapy arm.) N=42 subjects completed protocol therapy (n=23 in the intensive arm and n=19 in the standard arm.) All 42 that completed the study had platelet (PLT) measurements at both baseline and exit visits.
Measure: Mean (Standard Deviation); unit: *10^3 platelets/µL
Arm/Group | Stable Dosing | Intensive Dosing | Overall
Number analyzed (Participants) | 19 | 23 | 42
*10^3 platelets/µL | -10.92 (161.90) | -11.20 (145.78) | -11.07 (151.36)

21. Secondary Outcome: Median Change in Platelet Count (*10^3 Platelets/µL)
Description: as for outcome 8
Time Frame: From baseline at study entry to completion of therapy, up to 56 weeks
Population: as for outcome 20
Measure: Median (Full Range); unit: *10^3 platelets/µL
Arm/Group | Stable Dosing | Intensive Dosing | Overall
Number analyzed (Participants) | 19 | 23 | 42
*10^3 platelets/µL | -48 [-241 to 407] | -18 [-324 to 484] | -22 [-324 to 484]
Statistical Analysis 1: Comparison: Stable Dosing vs Intensive Dosing; Test type: Superiority; p = 0.75, Exact Wilcoxon (Mann-Whitney), two-sided

22. Secondary Outcome: Mean Change in Bilirubin (mg/dL)
Description: Descriptive statistics of the change between baseline and completion of the study will be provided.
Time Frame: From baseline at study entry to completion of therapy, up to 56 weeks
Population: Change calculations require subjects to have values at both baseline and exit visits. N=51 patients were randomized (n=25 to the Intensive arm and n=26 to the standard therapy arm.) N=42 subjects completed protocol therapy (n=23 in the intensive arm and n=19 in the standard arm.) Of the 42 that completed the study, n=40 had bilirubin measurements at both baseline and exit visits.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Stable Dosing | Intensive Dosing | Overall
Number analyzed (Participants) | 17 | 23 | 40
mg/dL | 0.24 (0.56) | -0.54 (1.05) | -0.21 (0.95)

23. Secondary Outcome: Median Change in Bilirubin (mg/dL)
Description: as for outcome 8
Time Frame: From baseline at study entry to completion of therapy, up to 56 weeks
Population: as for outcome 22
Measure: Median (Full Range); unit: mg/dL
Arm/Group | Stable Dosing | Intensive Dosing | Overall
Number analyzed (Participants) | 17 | 23 | 40
mg/dL | 0.30 [-0.80 to 1.30] | -0.30 [-4.60 to 1.00] | -0.07 [-4.60 to 1.30]
Statistical Analysis 1: Comparison: Stable Dosing vs Intensive Dosing; Test type: Superiority; p = 0.0013, Exact Wilcoxon (Mann-Whitney), two-sided

24. Secondary Outcome: Mean Change in Lactate Dehydrogenase (Units/L)
Description: as for outcome 8
Time Frame: From baseline at study entry to completion of therapy, up to 56 weeks
Population: Change calculations require subjects to have values at both baseline and exit visits. N=51 patients were randomized (n=25 to the Intensive arm and n=26 to the standard therapy arm.) N=42 subjects completed protocol therapy (n=23 in the intensive arm and n=19 in the standard arm.) Of the 42 that completed the study, n=41 had lactate dehydrogenase (LDH) measurements at both baseline and exit visits.
Measure: Mean (Standard Deviation); unit: units/L
Arm/Group | Stable Dosing | Intensive Dosing | Overall
Number analyzed (Participants) | 18 | 23 | 41
units/L | -11.94 (101.99) | -129.17 (181.47) | -77.71 (161.25)
Statistical Analysis 1: Comparison: Stable Dosing vs Intensive Dosing; Test type: Superiority; p = 0.013, t-test, 2 sided

25. Secondary Outcome: Median Change in Lactate Dehydrogenase (Units/L)
Description: Descriptive statistics of the change between baseline and completion of the study will be provided.
Time Frame: From baseline at study entry to completion of therapy, up to 56 weeks
Population: as for outcome 24
Measure: Median (Full Range); unit: units/L
Arm/Group | Stable Dosing | Intensive Dosing | Overall
Number analyzed (Participants) | 18 | 23 | 41
units/L | 4.5 [-189.0 to 219.0] | -94.0 [-477.0 to 248.0] | -54.0 [-477.0 to 248.0]

26. Secondary Outcome: Number of Participants Who do Not Have Normal Transcranial Doppler (TCD) Ultrasound Velocities
Description: Normal TCD velocities will be defined as TCD velocities <170 cm/s.
Time Frame: From baseline at study entry to completion of therapy, up to 56 weeks
Population: Subjects that complete protocol therapy and have TCD ultrasound at exit visit. N=42 subjects completed protocol therapy.
Measure: Count of Participants; unit: Participants
Arm/Group | Stable Dosing | Intensive Dosing
Number analyzed (Participants) | 5 | 6
Participants | 0 | 0

27. Secondary Outcome: Number of Participants Who Undergo Surgery
Description: Any operative procedure will be included.
Time Frame: From start of therapy through completion of therapy, up to 56 weeks
Population: Includes all randomized patients, n=51.
Measure: Count of Participants; unit: Participants
Arm/Group | Stable Dosing | Intensive Dosing
Number analyzed (Participants) | 26 | 25
Participants | 3 | 9

28. Secondary Outcome: Number of Participants Who Undergo Transfusion
Description: Transfusion will be defined as the provision of red blood cells to correct anemia.
Time Frame: From start of therapy through completion of therapy, up to 56 weeks
Population: Includes all randomized patients, n=51.
Measure: Count of Participants; unit: Participants
Arm/Group | Stable Dosing | Intensive Dosing
Number analyzed (Participants) | 26 | 25
Participants | 2 | 2

29. Secondary Outcome: Number of Patients With Toxicities Related to Hydroxyurea Dosing
Description: Number of patients with toxicities to include: neutropenia (ANC <1000*/µL), reticulocytopenia (ARC <80*10^3/µL and concomitant anemia (hemoglobin <6 g/dL), and thrombocytopenia (platelets <100*10^3/µL).
Time Frame: From start of therapy through completion of therapy, up to 56 weeks
Population: N=51 randomized patients (n=25 intensive arm and n=26 standard arm).
Measure: Count of Participants; unit: Participants
Arm/Group | Stable Dosing | Intensive Dosing
Number analyzed (Participants) | 26 | 25
Participants
  Neutropenia | 9 | 15
  Reticulocytopenia | 3 | 4
  Thrombocytopenia | 1 | 3
  Anemia | 0 | 0

30. Secondary Outcome: Number of Toxicities Related to Hydroxyurea Dosing
Description: Number of toxicities will be reported to include: neutropenia (ANC <1000*/µL), reticulocytopenia (ARC <80*10^3/µL and concomitant anemia (hemoglobin <6 g/dL), and thrombocytopenia (platelets <100*10^3/µL).
Time Frame: From start of therapy through completion of therapy, up to 56 weeks
Population: N=51 randomized patients (n=25 intensive arm and n=26 standard arm).
Measure: Number; unit: Toxicities
Arm/Group | Stable Dosing | Intensive Dosing
Number analyzed (Participants) | 26 | 25
Toxicities
  Neutropenia | 12 | 32
  Reticulocytopenia | 3 | 4
  Thrombocytopenia | 1 | 5
  Anemia | 0 | 0

31. Secondary Outcome: Change in Pain and Hurt Score
Description: Change in PedsQL 4.0 score will be reported. Scores are based on a 100 point scale, 0-100 with higher scores indicating a better quality of life. We are taking the exit visit score and subtracting the baseline score.
Time Frame: From baseline at study entry to completion of therapy, up to 56 weeks
Population: Of the N=51 randomized patients (n=25 intensive arm and n=26 standard arm), only 1 patient had The PedsQL ™ Sickle Cell Disease Module data at both baseline and exit visit.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Stable Dosing | Intensive Dosing
Number analyzed (Participants) | 1 | 0
score on a scale | 19.1 (NA) — Only 1 patient had data at both baseline and exit visit. |

32. Secondary Outcome: Change in Pain Impact Score
Description: as for outcome 31
Time Frame: From baseline at study entry to completion of therapy, up to 56 weeks
Population: as for outcome 31
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Stable Dosing | Intensive Dosing
Number analyzed (Participants) | 1 | 0
score on a scale | 15 (NA) — Only 1 patient had data at both baseline and exit visit. |

33. Secondary Outcome: Change in Pain Management Score
Description: as for outcome 31
Time Frame: From baseline at study entry to completion of therapy, up to 56 weeks
Population: as for outcome 31
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Stable Dosing | Intensive Dosing
Number analyzed (Participants) | 1 | 0
score on a scale | -25 (NA) — Only 1 patient had data at both baseline and exit visit. |

34. Secondary Outcome: Change in Worry I Score
Description: as for outcome 31
Time Frame: From baseline at study entry to completion of therapy, up to 56 weeks
Population: as for outcome 31
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Stable Dosing | Intensive Dosing
Number analyzed (Participants) | 1 | 0
score on a scale | 20 (NA) — Only 1 patient had data at both baseline and exit visit. |

35. Secondary Outcome: Change in Worry II Score
Description: as for outcome 31
Time Frame: From baseline at study entry to completion of therapy, up to 56 weeks
Population: as for outcome 31
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Stable Dosing | Intensive Dosing
Number analyzed (Participants) | 1 | 0
score on a scale | 20 (NA) — Only 1 patient had data at both baseline and exit visit. |

36. Secondary Outcome: Change in Emotions Score
Description: as for outcome 31
Time Frame: From baseline at study entry to completion of therapy, up to 56 weeks
Population: as for outcome 31
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Stable Dosing | Intensive Dosing
Number analyzed (Participants) | 1 | 0
score on a scale | 0 (NA) — Only 1 patient had data at both baseline and exit visit. |

37. Secondary Outcome: Change in Treatment Score
Description: as for outcome 31
Time Frame: From baseline at study entry to completion of therapy, up to 56 weeks
Population: as for outcome 31
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Stable Dosing | Intensive Dosing
Number analyzed (Participants) | 1 | 0
score on a scale | 37.5 (NA) — Only 1 patient had data at both baseline and exit visit. |

38. Secondary Outcome: Change in Communication I Score
Description: as for outcome 31
Time Frame: From baseline at study entry to completion of therapy, up to 56 weeks
Population: as for outcome 31
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Stable Dosing | Intensive Dosing
Number analyzed (Participants) | 1 | 0
score on a scale | 50 (NA) — Only 1 patient had data at both baseline and exit visit. |

39. Secondary Outcome: Change in Communication II Score
Description: as for outcome 31
Time Frame: From baseline at study entry to completion of therapy, up to 56 weeks
Population: as for outcome 31
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Stable Dosing | Intensive Dosing
Number analyzed (Participants) | 1 | 0
score on a scale | 8.3 (NA) — Only 1 patient had data at both baseline and exit visit. |

ADVERSE EVENTS:
Time Frame: Subjects in both treatment arms will be followed for a maximum of 56 weeks regardless of the actual number of study visits. Upon completion of the 56 weeks, patients will be followed for an additional 30 days for toxicities and will then be taken off study.
Groups:
- Stable Dosing - Post Randomization: In the first 8 weeks (± 2 weeks) of this study, participants will receive standard treatment [a fixed dose of 20 (± 2.5) mg/kg/day of hydroxyurea]. After 8 weeks (± 2 weeks) of standard treatment, participants will be randomized (like flipping a coin) to one of two treatment groups. Group 1 (Stable Dosing) continues standard treatment.
- Intensive Dosing - Post Randomization: In the first 8 weeks (± 2 weeks) of this study, participants will receive standard treatment [a fixed dose of 20 (± 2.5) mg/kg/day of hydroxyurea]. After 8 weeks (± 2 weeks) of standard treatment, participants will be randomized (like flipping a coin) to one of two treatment groups. Group 2 (Intensive Dosing) will have their HU dose increased by 5 mg/kg/day every 8 weeks up to a maximum of 35 mg/kg/day.
- All Participants - Pre Randomization: All participants enrolled
Arm/Group | Stable Dosing - Post Randomization | Intensive Dosing - Post Randomization | All Participants - Pre Randomization
All-Cause Mortality (participants affected / at risk) | 1/26 | 0/25 | 0/58
Serious Adverse Events (participants affected / at risk) | 3/26 | 2/25 | 1/58
Other Adverse Events (participants affected / at risk) | 2/26 | 8/25 | 3/58
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Stable Dosing - Post Randomization (N=26) | Intensive Dosing - Post Randomization (N=25) | All Participants - Pre Randomization (N=58)
Platelet count decreased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Immune system disorders,- Other specify (Immune system disorders) | 0 (0) | 0 (0) | 1 (1) — Fever in pediatric patient
Other (Specify_) (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) — "breath holding spell"
Neutropenia (Immune system disorders) | 0 (0) | 1 (1) | 0 (0)
Infections and infestations - Other, specify (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) — Norovirus/rotovirus diarrhea
Sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Surgical and medical procedures - Other specify (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) — Removal of foreign object
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Stable Dosing - Post Randomization (N=26) | Intensive Dosing - Post Randomization (N=25) | All Participants - Pre Randomization (N=58)
Febrile neutropenia (Blood and lymphatic system disorders) | 2 (2) | 6 (6) | 3 (3)
Platelet count decreased (Investigations) | 0 (0) | 2 (4) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-03-09): https://cdn.clinicaltrials.gov/large-docs/15/NCT03020615/Prot_SAP_000.pdf